CLINICAL TRIAL: NCT05848284
Title: Clinical Safety and Efficacy of the VDyne Transcatheter Tricuspid Valve Replacement System for the Treatment of Tricuspid Regurgitation
Brief Title: Clinical Safety and Efficacy of the VDyne Transcatheter Tricuspid Valve Replacement System for the Treatment of Tricuspid Regurgitation ( VISTA-US)
Acronym: VISTA-US
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VDyne, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TPR0037-P
Record Dates: First submitted 2023-03-29; First posted 2023-05-08 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Tricuspid Regurgitation; Tricuspid Valve Disease; Tricuspid Valvular Disorders
Keywords: VDyne
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- VDyne System Treatment Arm (Experimental): Device
  Interventions: Device: VDyne Transcatheter Tricuspid Valve Replacement System

INTERVENTIONS:
Device: VDyne Transcatheter Tricuspid Valve Replacement System — The study investigational device is the VDyne Transcatheter Tricuspid Valve Replacement System which consists of a bioprosthetic implantable tricuspid valve, the VDyne Delivery System, Drop Tether, accessories that facilitate the placement of the valve and the VDyne Retrieval System. The VDyne Valve is deployed by transfemoral implantation within the native tricuspid valve and is implanted under fluoroscopic and transesophageal echocardiography (TEE) guidance, while the heart remains beating, without the use of CPB. The valve is repositionable and fully retrievable intraoperatively. Repositioning allows optimization of the valve position following deployment, and retrieval, with the VDyne Retrieval System, allows use of an alternative valve size or removal of the index VDyne Valve in the event of suboptimal valve delivery or other intraoperative complication.
  Other Names: VDyne System; VDyne Tricuspid System; VDyne Valve System; VDyne Valve

SUMMARY:
The purpose of this clinical study is to evaluate the safety and clinical efficacy of the VDyne System in the treatment of symptomatic severe tricuspid regurgitation (TR).

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic severe tricuspid valve regurgitation of primary or secondary etiology.
* NYHA class ≥ II. If NYHA Class IV, patient must be ambulatory.
* Subject is adequately treated with medical therapy for heart failure ≥ 30 days prior to
* index procedure, including a diuretic.
* Heart Team determines patient is a recommended candidate for the VDyne System.
* Age >18 years at time of index procedure.
* Clinical Screening Committee (CSC) and Imaging Core Labs confirm suitability for treatment with the VDyne System.

Exclusion Criteria:

* Patient anatomy (cardiac and vascular) is not suitable for VDyne System as assessed by Imaging Core Labs, Sponsor or Clinical Screening Committee (CSC)
* Intolerance to procedural anticoagulation or post-procedural antiplatelet/ anticoagulation regimen that cannot be medically managed
* Hypersensitivity to nickel or titanium
* Left Ventricular Ejection Fraction (LVEF) <30%.
* Severe RV dysfunction.
* Significant abnormalities of the tricuspid valve and sub-valvular apparatus.
* Sepsis including active infective endocarditis (IE) (within last 6 months).
* Right ventricular, atrial thrombus, vegetation or mass on tricuspid valve.
* Severe tricuspid annular or leaflets calcification.
* Systolic pulmonary hypertension with systolic pulmonary artery pressure >70 mmHg.
* History or rheumatic fever
* Significant coronary artery disease requiring treatment such as symptomatic, unresolved multi-vessel or unprotected left main coronary artery disease.
* Any planned surgery or interventional procedure within 30 days prior to or 30 days following the implant procedure. This includes any planned concomitant cardiovascular procedure such as CABG, PCI, pulmonary vein ablation, left atrial appendage occlusion, septal defect repair, etc.
* Unresolved severe symptomatic carotid stenosis (> 70% by ultrasound).
* Cardiac resynchronization therapy device or implantable pulse generator implanted within 60 days of planned implant procedure.
* Permanent pacing leads that will interfere with delivery or implantation of the VDyne Valve.
* Cardiogenic shock or hemodynamic instability requiring inotropes or mechanical support devices at the time of planned implant procedure.
* Prior tricuspid valve surgery or catheter-based therapy with permanent residual device(s) implanted that would preclude delivery or implantation of the VDyne Valve (e.g. valve replacement, edge to edge repair, etc.).
* Significant valvular heart disease requiring intervention other than the tricuspid valve.
* Known significant intracardiac shunt (e.g. septal defect)
* Cerebrovascular accident (stroke, TIA) within 6 months of treatment procedure.
* Severe lung disease (severe COPD or continuous use of home oxygen or oral steroids).
* Acute myocardial infarction (AMI) within 30 days.
* Significant renal dysfunction (eGFR<30 ml/min/1.73m2) or on dialysis.
* End-stage liver disease (MELD > 11 / CHILD class C).
* Bleeding requiring transfusion within prior 30 days.
* Coagulopathy or other clotting disorder that cannot be medically managed.
* Chronic immunosuppression or other condition that could impair healing response.
* Any of the following: leukopenia, chronic anemia (Hgb < 9), thrombocytopenia, history of bleeding diathesis, or coagulopathy.
* Unwilling to receive blood products.
* Known hypersensitivity or contraindication to procedural or post-procedural medications (e.g., contrast solution) which cannot be adequately managed medically.
* Life expectancy less than 12 months due to non-cardiac comorbidities.
* Treatment is not expected to provide benefit (futile).
* Current IV Drug user (must be free drug abuse for > 1 year).
* Pregnant, lactating or planning pregnancy within next 12 months.
* Vulnerable patient groups (minors, cognitively impaired persons, prisoners, persons whose willingness to volunteer could be unduly influenced by the expectation of benefits associated with participation or of retaliatory response from senior members of a hierarchy in case of refusal to participate, such as students, residents, and employees).
* Currently participating in an investigational drug or device trial that has not reached its primary endpoint or is likely to interfere with this study.
* Patient (or legal guardian) unable or unwilling to provide written, informed consent before study enrollment.
* Patient unable or unwilling to comply with study required testing and follow-up visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2030-11-30 (Estimated)

PRIMARY OUTCOMES:
The percentage of subjects with Device- and/or Procedure-related Major Adverse Events (MAE) within 30 days of the procedure, as classified by the Clinical Events Committee (CEC). | Implant to 30 days post-procedure
  The percentage of subjects with Device- and/or Procedure-related Major Adverse Events (MAE) within 30 days of the procedure, as classified by the Clinical Events Committee (CEC).
Change in tricuspid valve regurgitation compared to baseline as measured by the Imaging Core Labs | Baseline to 1 month after implant
  Change in tricuspid valve regurgitation compared to baseline as measured by the Imaging Core Labs
Changes in symptom status (NYHA class) | Baseline to 1 month after implant
  Changes in symptom status (NYHA class)
Changes in functional capacity (6-minute walk test) | Baseline to 1 month after implant
  Changes in functional capacity (6-minute walk test)
Changes in in quality of life (KCCQ score) | Baseline to 1 month after implant
  Changes in in quality of life (KCCQ score). A higher score indicates worsening quality of life outcomes

SECONDARY OUTCOMES:
The percentage of subjects with Device- and/or Procedure-related Major Adverse Events (MAE) after 30 days to 1 year of the procedure, as classified by the Clinical Events Committee (CEC). | 30 days post-procedure to 1 year
  The percentage of subjects with Device- and/or Procedure-related Major Adverse Events (MAE) after 30 days to 1 year of the procedure, as classified by the Clinical Events Committee (CEC).
Change in tricuspid valve regurgitation compared to baseline as measured by the Imaging Core Labs | 1 month after implant to 1 year post-implant
  Change in tricuspid valve regurgitation compared to baseline as measured by the Imaging Core Labs
Changes in right ventricle as measured by core lab | 1 month after implant to 1 year post-implant
  Changes in the right ventricle as measured by core lab
Rate of heart failure hospitalization | 1 month after implant to 1 year post-implant
  Rate of heart failure hospitalization
Changes in symptom status (NYHA class) | 1 month after implant to 1 year post-implant
  Changes in symptom status (NYHA class)
Changes in functional capacity (6-minute walk test) | 1 month after implant to 1 year post-implant
  Changes in functional capacity (6-minute walk test)
Changes in in quality of life (KCCQ score). | 1 month after implant to 1 year post-implant
  Changes in in quality of life (KCCQ score). A higher score indicates worsening outcomes

CONTACTS AND LOCATIONS:
Locations (11):
- United States (10):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Los Robles Hospital and Medical Center, Thousand Oaks, California
  - Henry Ford Hospital, Detriot, Michigan
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Columbia University Medical Center/NYPH, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Oregon Health and Science Unversity, Portland, Oregon
  - Medical University of South Carolina, Charleston, South Carolina
  - Ascension St. Thomas, Nashville, Tennessee
- Québec-Université Laval (IUCPQ-ULaval), Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://www.vdyne.com